CLINICAL TRIAL: NCT00296153
Title: Omacor; Omega-3-Acid Ethyl Ester 90 (n-3 PUFA) and Risk Factors in HIV Infected Patients Treated With HAART, With Special Focus on Lipids
Brief Title: Omacor and Cardiovascular Risk Factors in HIV Patients on HAART Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Runar Vige, Pronova BioPharma
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTN K85 05026; Eudract no: 2005-005135-10
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Human Immunodeficiency Virus; Ischemic Heart Disease
Keywords: Human immunodeficiency Virus (HIV); Highly Active Antiviral Therapy (HAART); Ischemic Heart Disease; OMACOR; Triglycerides; Endothelial function; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Omacor 1000mg x 4 / day
  Interventions: Drug: Omega-3-acid ethyl esters 90
- 2 (Placebo Comparator)
  Interventions: Drug: Omega-3-acid ethyl esters 90

INTERVENTIONS:
Drug: Omega-3-acid ethyl esters 90 — Omacor capsule 1000mg x 4 per day. Duration 12 weeks
  Other Names: Omacor versus placebo

SUMMARY:
The purpose of this study is to evaluate the effect of Omacor 4g/day on blood lipid parameters and on the function and stiffness of blood vessels in HIV infected patients on Antiretroviral Therapy (HAART)

DETAILED DESCRIPTION:
Results from recent studies show increasing numbers of Ischemic Heart Disease (IHD) incidents among patients on HAART treatment (Highly Active Antiviral Therapy). Three elements have received special attention:

1. the immunodeficient effects of the HIV infection itself may influence the progression of arteriosclerosis
2. the higher levels of risk behaviour in this group of patients (i.e. high prevalence of smokers in this group)
3. The HAART treatment itself increases plasma levels of cholesterol, LDL cholesterol and triglycerides, resulting in HIV related lipodystrophy.

The cardioprotective effects of n-3 PUFAs are well established both through epidemiological studies and through small and large clinical trials. Clinical trials have shown positive effects of n-3 PUFA on plasma triglycerides, and statistically significant reductions in cardiovascular death and sudden cardiac death. Moreover n-3 PUFAs have been shown to have beneficial effects on endothelial function. Based on the above rationale it is expected that Omacor (Omega-3-acid ethyl ester 90) will have positive effects on risk factors related to Ischemic Heart Disease in HIV patients on HAART treatment.

Approximately 50 patients will be randomized to Omacor 4 grams/day or placebo. Treatment period is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Man/women > 18 years of age
* Documented HIV infection
* On active treatment with HAART for at least 3 months.
* Written informed consent. This implies that the patient can read and understand Danish or English

Exclusion Criteria:

* Age < 18 years
* Malign disease
* Patients assessed as not cooperative
* Patients planning to be pregnant or who are already pregnant or breast feeding.
* Patients who have been taking fish oil capsules prior to randomization. However, patients who have discontinued fish oil supplements at least 8 weeks prior to the first visit will be included
* Patients allergic to fish proteins
* Statin treatment that has been ongoing for less than three months, or a change in statin treatment dose within the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The change from week 0 (baseline) to week 12 for: Plasma triglycerides | baseline and 12 weeks

SECONDARY OUTCOMES:
The change from week 0 (baseline) to week 12 for: Pulse Wave Velocity, Flow medicated vasodilation | baseline and 12 weeks
HDL-cholesterol, LDL-cholesterol, total cholesterol | baseline and 12 weeks
Inflammatory parameters: ICAM, VCAM, sensitive CRP | baseline and 12 weeks
Apo A, Apo B, Lp(a), fibrinogen, PAI-1 ag, vw-Factor, thrombomodulin, oxidized LDL, small dense LDL, LTB4 from stimulated granulocytes | baseline and 12 weeks
Safety parameters | baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe H. Christensen, PhD, Principal Investigator — Aalborg Hospital, Department of Nephrology
Locations (1):
- Aalborg Hospital, Department of Nephrology, Aalborg, Denmark